CLINICAL TRIAL: NCT07013474
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 3, RANDOMIZED, DOUBLE-BLIND, 3-ARM STUDY TO INVESTIGATE IBUZATRELVIR IN ADULTS WITH SYMPTOMATIC COVID-19 WHO ARE SEVERELY IMMUNOCOMPROMISED
Brief Title: A Study to Learn About the Study Medicine Ibuzatrelvir in Adults With COVID-19 Who Are Severely Immunocompromised
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C5091018; 2024-517671-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-05-05; First posted 2025-06-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: COVID-19 Infection
Keywords: COVID-19 infection; pneumonia; respiratory tract infections; coronavirus infection; RNA virus infection; lung disease; pneumonia, viral; infections; virus; viral protease inhibitor; protease inhibitor; enzyme inhibitor; severe immunocompromise; anti-viral agents; anti-infectives; ibuzatrelvir; remdesivir; COVID-19
MeSH Terms: conditions — COVID-19; Pneumonia; Respiratory Tract Infections; Coronavirus Infections; RNA Virus Infections; Lung Diseases; Pneumonia, Viral; Infections; Virus Diseases | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, with required dedicated unblinded staff for dose preparation for remdesivir and placebo for remdesivir.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ibuzatrelvir (Experimental): Participants will receive ibuzatrelvir orally twice a day + IV placebo for remdesivir
  Interventions: Drug: ibuzatrelvir; Drug: placebo for remdesivir
- Ibuzatrelvir + Remdesivir (Experimental): Participants will receive ibuzatrelvir orally twice a day + IV remdesivir
  Interventions: Drug: ibuzatrelvir; Drug: remdesivir
- Remdesivir (Experimental): Participants will receive placebo for ibuzatrelvir orally twice a day + IV remdesivir
  Interventions: Drug: remdesivir; Drug: placebo for ibuzatrelvir

INTERVENTIONS:
Drug: ibuzatrelvir — tablet
  Arms: Ibuzatrelvir; Ibuzatrelvir + Remdesivir
Drug: remdesivir — injection, for intravenous use
  Other Names: veklury
  Arms: Ibuzatrelvir + Remdesivir; Remdesivir
Drug: placebo for ibuzatrelvir — tablet
  Arms: Remdesivir
Drug: placebo for remdesivir — injection, for intravenous use
  Arms: Ibuzatrelvir

SUMMARY:
This is a Phase 3, randomized, actively controlled, double-blinded, double-dummy, superiority study to evaluate the efficacy and safety of ibuzatrelvir alone and in combination with remdesivir IV compared to remdesivir IV alone for the treatment of symptomatic COVID-19 in severely immunocompromised adult participants who are non-hospitalized or are hospitalized for observation or study intervention administration but do not require supplemental oxygen for COVID-19.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to learn about a study medicine called Ibuzatrelvir for the possible treatment of COVID-19 in immunocompromised patients. Immunocompromised patients with COVID-19 have more difficulty fighting infections and are at risk for persistent infections and progression to severe illness. This patient population may benefit from extended antiviral treatment durations, or a combination of antiviral therapies. This study will evaluate the efficacy and safety of ibuzatrelvir with and without remdesivir compared with remdesivir alone for the treatment of symptomatic COVID-19 in adult participants who are severely immunocompromised.

The study is seeking adult male and female participants who:

* Have a confirmed COVID-19 infection
* Are severely immunocompromised due to blood cancers, organ transplant, certain medications or therapies
* Have experienced the onset of signs or symptoms of COVID-19 within the past 5 days and are currently experiencing at least one of them.

All of the participants in this study will receive active treatment for COVID-19, and will be randomized to one of three treatment arms. One-third will received remdesivir, one-third will receive ibuzatrelvir, and one third will receive both remdesivir and ibuzatrelvir. Ibuzatrelvir will be taken by mouth twice daily, and remdesivir is given as an IV infusion daily. Placebos that look like the study medicines but do not have any medication will be given to make the 3 treatment arms appear to be the same. The study will compare the experiences of people receiving ibuzatrelvir with and without remdesivir to those of the people who only received remdesivir for COVID-19. This will help decide if ibuzatrelvir is safe and effective.

Participants will attend about 10 study visits over 24 weeks. During this time, they will have:

* visits at the study clinic
* blood work
* swabs of the nose that are collected in the clinic and also by participants at home
* questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older at screening who are non-hospitalized or hospitalized for observation or with the intent of administering the study intervention.
2. Confirmed SARS-CoV-2 infection as determined by RAT (or other locally approved test) collected within 2 days prior to randomization. Initial onset of symptoms attributable to COVID-19 within 5 days prior to the day of randomization and at least 1 of the specified symptoms attributable to COVID-19 present on the day of randomization.
3. Severely immunocompromised due to:

   * Solid organ or islet cell transplant recipient who is receiving immunosuppressive therapy;
   * Active hematologic malignancy (eg, chronic lymphocytic leukemia, non-Hodgkin lymphoma, multiple myeloma, acute leukemia);
   * Receipt of CAR-T-cell therapy or HCT either within 2 years of transplantation or who are receiving immunosuppressive therapy;
   * Currently receiving or recently received B-cell depleting therapies (eg, rituximab), where the immunosuppressive effect is still ongoing.

Exclusion Criteria:

1. Severe COVID-19, or current need for supplemental oxygen for treatment of COVID-19.
2. Receiving dialysis or have current kidney failure (ie, eGFR consistently <15 mL/min/1.73 m2)
3. Active liver disease
4. History of hypersensitivity or other contraindication to any of the components of the study interventions, as determined by the investigator
5. Suspected or confirmed concurrent active systemic infection other than COVID-19 that may interfere with the evaluation of response to the study intervention.
6. Life expectancy less than 30 days at study entry due to an underlying condition, in the judgement of the investigator.
7. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Has received any other antiviral for the treatment of the current COVID-19 infection
9. Current use of any prohibited concomitant medication(s) or unwillingness or inability to use a required concomitant medication(s).
10. Current or previous administration of an investigational product (drug or vaccine) within 30 days (or as determined by local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer). Authorized or products with conditional approval are not considered investigational.
11. Prior participation in this trial or any clinical trial of ibuzatrelvir.
12. Females who are pregnant, breastfeeding, or who are planning to become pregnant within the timeframe of the study.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of patients meeting the primary composite endpoint, between ibuzatrelvir and remdesivir vs remdesivir groups in symptomatic adult participants with COVID-19 who are severely immunocompromised | 38 days
  The difference in the proportion of participants with the composite endpoint of a) COVID-19-related ED visits with administration of supplemental oxygen, COVID-19 antiviral, or IV treatment; COVID-19-related hospitalization; or all-cause mortality, and b) Evidence of recurrent or persistent SARS-CoV-2 infection

SECONDARY OUTCOMES:
Time to sustained alleviation of all targeted COVID-19 symptoms | 38 days
  The difference in median time to sustained alleviation of all targeted symptoms. Symptoms will be assessed through a daily electronic diary and include sore throat, cough, fever and diarrhea, among others.
Proportion of participants with evidence of recurrent or persistent SARS-CoV-2 infection. | 38 days
  The viral load is measured in nasal or nasopharyngeal samples using reverse transcription polymerase chain reaction (RT-PCR)
Proportion of participants with COVID-19-related ED visits with administration of supplemental oxygen, COVID-19 antiviral, or IV treatment, COVID-19-related hospitalization, or all-cause mortality. | 38 days
  Proportion of participants with COVID-19-related ED visits with administration of supplemental oxygen, COVID-19 antiviral, or IV treatment (eg, hydration, antibiotics, or corticosteroids), COVID-19-related hospitalization, or all-cause mortality.
Change from baseline in SARS-CoV-2 RNA level in NP or nasal swabs over time | 38 days
  The viral load is measured in nasal or nasopharyngeal samples using reverse transcription polymerase chain reaction (RT-PCR)
Proportion of participants with SARS-CoV-2 NP or nasal RNA <LLOQ at each time point | 38 days
  Proportion of participants with a SARS-CoV-2 viral load below the lower limit of quantification (LLOQ) of the assay used to measure it.
Proportion of participants with viral rebound in SARS-CoV-2 RNA level in NP or nasal swabs | 38 days
  Virologic rebound is defined as:
  * Viral RNA is not detectable at the end of treatment, and later is detectable through Day 38
  * Viral RNA is detected at end of treatment, and viral RNA levels increase further through Day 38
Time to sustained NP or nasal swab SARS-CoV-2 RNA <LLOQ | 38 days
  The time it takes for the viral RNA to no longer be detectable in a sample
Incidence of Treatment emergent adverse events, serious adverse events, and adverse events leading to discontinuation | 38 days
  An adverse event (AE) is any untoward medical occurrence in a participant, temporarily associated with the use of study intervention, whether or not considered related to the study intervention. Serious adverse event (SAE) is any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/ incapacity; congenital anomaly/birth defect; a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical events. AEs included both SAEs and all non-SAEs. An AE is considered as TEAE if the event started on or after start date of study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (114):
- United States (46):
  - Hope Clinical Research, Inc., Canoga Park, California
  - Amicis Research Center - Granada Hills, Granada Hills, California
  - UC Davis CTSC Clinical Research Center, Sacramento, California
  - University of California Davis Health, Sacramento, California
  - UCHealth Anschutz Inpatient Pavilion - Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Clinical and Translational Research Center, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - BRP- Hialeah Hospital, Hialeah, Florida
  - D&H Cancer Research Center LLC, Margate, Florida
  - Kendall South Medical Center, Miami, Florida
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Humphreys Diabetes Center, Boise, Idaho
  - St. Luke's Idaho Elks Children's Pavilion, Boise, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Trials Center, Boston, Massachusetts
  - Clinical Trials Hub, Boston, Massachusetts
  - Skylight Health Research - Burlington, Burlington, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Profound Research LLC, Farmington Hills, Michigan
  - Revive Research Institute, Inc., Farmington Hills, Michigan
  - Holy Name Medical Center, Teaneck, New Jersey
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Duke Main Hospital and Clinics, Durham, North Carolina
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Cincinnati College of Medicine (UC Holmes), Cincinnati, Ohio
  - West Tennessee Research Institute, Jackson, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UT Physicians, Houston, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
  - Swedish Ambulatory Infusion Center- First Hill, Seattle, Washington
  - Swedish Cancer Institute Treatment Center, Seattle, Washington
  - Swedish Medical Center- Innovative Therapeutics & Research Unit, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - Swedish Medical Center - First Hill Campus, Seattle, Washington
- Belgium (4):
  - UZ Brussel, Brussels, Brussels Capital
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-capitale, Région de
  - AZ Sint-Jan Brugge-Oostende AV, Bruges, West-vlaanderen
  - Jules Bordet Institute, Anderlecht
- Brazil (5):
  - School of Medicine Federal University of Minas Gerais, Belo Horizonte, Minas Gerais
  - Unidade de Pesquisa Clínica em Vacinas da Faculdade de Medicina da Universidade Federal de Minas Ger, Belo Horizonte, Minas Gerais
  - Hospital de Clinicas de Porto Alegre, Bairro Santa Cecília, Rio Grande do Sul
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
- Denmark (4):
  - Rigshospitalet, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
  - Odense Universitetshospital, Odense, Region Syddanmark
- France (5):
  - Hopital Claude Huriez - CHU de Lille, Lille, NORD
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Hôpital Saint Antoine, Paris
  - Hôpital Bichat - Claude-Bernard, Paris
  - Hôpital Saint-Louis, Paris, Île-de-France Region
- Germany (2):
  - TUM Klinikum, München, Bavaria
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
- Greece (4):
  - University General Hospital of Alexandroupoli, Alexandroupoli, Anatolikí Makedonía KAI Thráki
  - Evangelismos General Hospital of Athens, Athens, Attikí
  - Alexandra General Hospital of Athens, Athens, Attikí
  - General Hospital of Athens "Laiko", Athens, Attikí
- Japan (10):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Rinku General Medical Center, Izumisano, Osaka
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - National Center for Global Health and Medicine, Shinjuku, Tokyo
  - Tachikawa Hospital, Tachikawa, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Nagasaki University Hospital, Nagasaki
  - Saga University Hospital, Saga
- Radboudumc, Nijmegen, Netherlands
- Puerto Rico (2):
  - BRCR Medical Center - Ponce, Ponce
  - BRCR Global Puerto Rico, San Juan
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica, Banská Bystrica Region
  - Narodny ustav detskych chorob, Bratislava, Bratislava Region
  - Fakultna nemocnica Trnava, Trnava, Trnava Region
  - Narodny onkologicky ustav, Bratislava
  - Nemocnica s poliklinikou Stefana Kukuru Michalovce, a.s., Michalovce
- South Korea (4):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - Chonnam National University Hospital, Gwangju, Kwangju-kwangyǒkshi
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (10):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - CHUVI- Hospital Alvaro Cunqueiro, Vigo, Pontevedra [pontevedra]
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Virgen de Valme, Seville
- Karolinska Universitetssjukhuset Huddinge, Huddinge, Sweden
- Taiwan (4):
  - Far Eastern Memorial Hospital, New Taipei City, NEW Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (7):
  - Acibadem Universitesi Atakent Hastanesi, Istanbul, İ̇stanbul
  - Hacettepe Universite Hastaneleri, Ankara
  - Ibni Sina Hospital, Ankara
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Kocaeli Üniversitesi, Kocaeli
  - Sakarya Training and Research Hospital, Sakarya
  - Karadeniz Technical University, Trabzon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091018
- See also: Pfizer Clinical Trials website — https://www.pfizerclinicaltrials.com/nct07013474-covid-19-trial